CLINICAL TRIAL: NCT00755586
Title: Autologous Bone Marrow Transplantation for Muscle Improvement in Traumatic Brachial Plexus Injuries
Brief Title: Stem Cell Therapy to Improve the Muscle Function of Patients With Partly Denervated Muscles of the Arm
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Prof.dr. R.G.H.H. Nelissen, Leiden University Medical Center, department of orthopaedics
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40-41200-98-040
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Brachial Plexus Injury
Keywords: Brachial plexus; Muscle denervation; Stem cell transplantation; Bone marrow cells; Satellite cells; Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Procedure: Mononuclear cell injection: 4 * 10e8 cells
- B (Experimental)
  Interventions: Procedure: Mononuclear cell injection: 8 * 10e8 cells
- C (No Intervention)
  Interventions: Procedure: No mononuclear cell injection

INTERVENTIONS:
Procedure: Mononuclear cell injection: 4 * 10e8 cells — 350 ml bone marrow will be aspirated from the posterior iliac crest under general anesthesia in combination with a muscle tendon transposition surgery. Next, the patients will receive a bone marrow derived mononuclear cell injection of 4 * 10e8 cells in the m. biceps brachii.
  Arms: A
Procedure: Mononuclear cell injection: 8 * 10e8 cells — 650 ml bone marrow will be aspirated from the posterior iliac crest under general anesthesia in combination with a muscle tendon transposition surgery. Next, the patients will receive a bone marrow derived mononuclear cell injection of 8 * 10e8 cells in the m. biceps brachii.
  Arms: B
Procedure: No mononuclear cell injection — Patients will receive a muscle tendon transposition surgery without bone marrow aspiration or mononuclear cell injection.
  Arms: C

SUMMARY:
The purpose of this study is to assess muscle improvement after stem cell injection in the biceps muscle of patients with a brachial plexus injury.

DETAILED DESCRIPTION:
Brachial plexus injuries can cause severe disabilities and often affect young adults and newborn children. When initial conservative treatment or nerve surgery fails, muscle/tendon transfers are the only current treatment options available to regain a functional arm. During this extensive surgery a healthy donor muscle is transposed to exert a different function. After long-term denervation the muscle is irreversibly changed. Muscle atrophy, fattening, fibrosis, decrease in capillary to muscle fiber ratio and decline in the number of satellite cells, which are responsible for post-natal muscle repair, is seen. For neuromuscular diseases, cell therapy aiming at rescuing muscle damage by delivery of cells that can differentiate into skeletal muscle, might be a promising approach. Safety questions remain whether stem cell injection results in non-muscle tissue formation like inflammatory cells or connective tissue formation in the transplanted muscles. Furthermore, it remains to be determined whether these stem cells undergo functional integration and enhance muscle function. The objective of this pilot study is to assess functional and morphological improvement of the m. biceps brachii after autologous bone marrow-derived mononuclear cell injection.

ELIGIBILITY:
Inclusion Criteria:

* BP patients with paresis of m. biceps brachii (MRC 1,2,3), either after conservative treatment or at least two years after nerve surgery with partial recovery of the elbow flexor
* Patients capable and willing to give informed consent

Exclusion Criteria:

* Function recovery of the elbow flexor (m. biceps brachii) to a MRC motor scale of 0
* EMG activity: no motor unit potentials
* Medical history of other central of peripheral neurological disorders
* Inability to undergo BM harvesting
* Bleeding diathesis, INR > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
To assess muscle improvement, muscle biopsies, quantitative needle EMGs, muscle density analysis, force measurement, range of motion of the elbow joint and quality of life questionnaires will be performed. | Two years

SECONDARY OUTCOMES:
The secondary research aim of this study is to assess vital signs and to detect signs of hematoma and/or injection at the bone marrow aspiration site, injection site and/or surgical wound. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Rob GHH Nelissen, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands